CLINICAL TRIAL: NCT06460779
Title: Association of Age, Gross Motor Function With Activities of Daily Living, Participation in Home and Community in Children With Cerebral Palsy
Brief Title: Gross Motor Function and Living Skills in CP
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0792
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; childhood disablity; gross and motor function; participation; quality of life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) is non-progressive disorder, which undergoes mishap to the developing brain and it affects a person's ability to move and maintain balance and posture. Old name of CP is "Little's disease".Through social and community participation, children and youth with cerebral palsy (CP) form friendships, gain knowledge, learn skills, express creativity, and determine meaning and purpose in life. The purpose of this study is (1) to determine whether social and community participation of children and youth with CP differ based on age, sex, and gross motor function, and (2) to identify the types of activities in which social and community participation are highest

DETAILED DESCRIPTION:
Those participants will be excluded having any unstable medical condition that precluded safe community physical activity, any orthopedic or neurological surgery in the previous 6 months, moderate to profound intellectual disability, moderate to severe communication disability, severe visual impairment, any sensory impairment or psychological disorder. The tools that will be used are WHODAS 2.0(WHO Disability Assessment Schedule), Washington Group Short Set of Disability Questions, Child and Adolescent Scale of Participation Activities of Daily Living, Functional Mobility and Participation. Data will be analyzed on SPSS version 25, normality of the data will be checked and data will be presented in the form of descriptive statistics, mean, SD range correlation.

ELIGIBILITY:
Inclusion Criteria:

Washington Group on Disability Statistics (WG) score greater than or equal to 12.

* Children with age group of 6 to 12 years.
* With diagnosis of CP.
* WHOdas Cognition - score 2.5.
* Mobility - score 2.5.
* Self-care - score 2.5 attending to one's hygiene, dressing, eating and staying alone.
* Getting along -score 2.5 interacting with other people.
* Life activities -score 2.5 domestic responsibilities, leisure, work and school.
* Participation - score 2.5 joining in community activities, participating in society

Exclusion Criteria:

Any unstable medical condition that precluded safe community physical activity.

* Having any orthopedic or neurological surgery in the previous 6 months.
* Moderate to profound Intellectual disability.
* Moderate to severe communication disability.
* Severe visual impairmen

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: we measure age, gross motor function. ADLS in CP with the sample size of 100 students of schools under age 6-12 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Washington Group Short Set of Disability Questions | 6 weeks
  The WG-SS is intended for use in censuses and surveys To maximize international comparability, the WG-SS obtains information on difficulties a person may have in undertaking basic functioning activities that apply to people in all cultures and societies and of all nationalities and so are universally applicable.
Child and Adolescent Scale of Participation | 6 weeks
  The CASP is a 20-items 4-scales parent-report instrument covering attendance and involvement in the areas "home", "community", "school", and "living activities".
Communication Function Classification System | 6 weeks
  The CFCS is a tool used to classify the everyday communication of an individual with cerebral palsy into one of five levels according to effectiveness of communication. It consists of five levels which describe everyday communication ability

SECONDARY OUTCOMES:
WHODAS 2.0 participation in home and community in children with cerebral palsy | 6 weeks
  practical, generic assessment instrument that can measure health and disability at population level. It captures the level of functioning in 6 domains of life

CONTACTS AND LOCATIONS:
Overall Officials: saman ali, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colver A, McConachie H, Le Couteur A, Dovey-Pearce G, Mann KD, McDonagh JE, Pearce MS, Vale L, Merrick H, Parr JR; Transition Collaborative Group. A longitudinal, observational study of the features of transitional healthcare associated with better outcomes for young people with long-term conditions. BMC Med. 2018 Jul 23;16(1):111. doi: 10.1186/s12916-018-1102-y. PMID 30032726
- [Background] Liao YT, Hwang AW, Liao HF, Granlund M, Kang LJ. Understanding the Participation in Home, School, and Community Activities Reported by Children with Disabilities and Their Parents: A Pilot Study. Int J Environ Res Public Health. 2019 Jun 24;16(12):2217. doi: 10.3390/ijerph16122217. PMID 31238490